CLINICAL TRIAL: NCT01892345
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Trial to Evaluate the Safety and Efficacy of Eculizumab in Patients With Relapsing Neuromyelitis Optica (NMO)
Brief Title: A Randomized Controlled Trial of Eculizumab in AQP4 Antibody-positive Participants With NMO (PREVENT Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECU-NMO-301
Record Dates: First submitted 2013-06-20; First posted 2013-07-04 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Devic's disease, Transverse Myelitis; Optic Neuritis; relapse; eculizumab; soliris; NMO-IgG; CNS Autoimmune Disorders; Demyelinating Disorders; NMO; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis; Recurrence; Demyelinating Diseases | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eculizumab (Experimental): Biological/Vaccine: Eculizumab; Induction Period: Participants received eculizumab (900 milligrams [mg]) via intravenous (IV) infusion once a week (every 7 ± 2 days) for 4 weeks followed by eculizumab 1200 mg for the fifth dose (Week 4). This was followed by the Maintenance Period: Participants received eculizumab (1200 mg) via IV infusion every 2 weeks (every 14 ± 2 days) from the sixth dose (Week 6) onwards.
  Interventions: Drug: Eculizumab
- Placebo (Placebo Comparator): Placebo contains the same buffer components without the active ingredient. Induction Period: Participants received matching placebo (900 mg) via IV infusion once a week (every 7 ± 2 days) for 4 weeks, followed by matching placebo (1200 mg) for the fifth dose (Week 4). This was followed by the Maintenance Period: Participants received matching placebo (1200 mg) via IV infusion every 2 weeks (every 14 ± 2 days) from the sixth dose (Week 6) onwards.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eculizumab — Induction Phase: 900 mg IV weekly for 4 weeks, followed by 1200 mg for the fifth dose; Maintenance Phase: 1200 mg IV every 2 weeks
  Other Names: Soliris
  Arms: Eculizumab
Drug: Placebo — Induction Phase: matching placebo (900 mg) IV weekly for 4 weeks, followed by matching placebo (1200 mg) for the fifth dose; Maintenance Phase: matching placebo (1200 mg) IV every 2 weeks
  Arms: Placebo

SUMMARY:
The objectives of this time-to-event study were to assess the efficacy and safety of eculizumab as compared with placebo in participants with neuromyelitis optica spectrum disorder (NMOSD) who were anti-aquaporin-4 (AQP4) antibody-positive.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants ≥ 18 years old.
2. Diagnosis of NMO or NMOSD.
3. AQP4 antibody seropositive.
4. Historical relapse of at least 2 relapses in the last 12 months or 3 relapses in the last 24 months with at least 1 relapse in the 12 months prior to the screening.
5. Expanded Disability Status Scale score ≤ 7.
6. If a participant entered the study receiving immunosuppressive therapy (IST) for relapse prevention, the participant must have been on a stable maintenance dose of IST(s), as defined by the treating physician, prior to Screening and must have remained on that dose for the duration of the study, unless the participant experienced a relapse.
7. Female participants of childbearing potential were to have a negative pregnancy test (serum human chorionic gonadotropin). Participants were required to practice an effective, reliable, and medically approved contraceptive regimen during the study and for up to 5 months following discontinuation of treatment.

Key Exclusion Criteria:

1. Use of rituximab within 3 months prior to Screening.
2. Use of mitoxantrone within 3 months prior to Screening.
3. Use of intravenous immunoglobulin within 3 weeks prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (70):
- United States (19):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The Research Center of Southern California, Carlsbad, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami McKnight Brain Institute, Miami, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Multiple Sclerosis Comprehensive Care Center, NYU Langone Medical Center, New York, New York
  - The Ohio State University, Wexner Medical Center, CarePoint at Gahanna, Gahanna, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Multiple Sclerosis Treatment Center of Dallas, Dallas, Texas
  - University of Utah Health Care, Salt Lake City, Utah
  - Swedish Neuroscience Institute, Seattle, Washington
- Argentina (4):
  - Hospital General de Agudos Juan Antonio Fernandez, Ciudad Autonoma, Buenos Aires, Buenos Aires
  - Hospital J. M. Ramos Mejia, Ciudad Autonoma, Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Fundacion Rosarina de Neuro Rehabilitacion, Rosario, Santa Fe Province
- Australia (2):
  - University of Sydney, Brain and Mind Center, Camperdown, New South Wales
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Vseobecna fakultni nemocnice Neurologicka klinika, Prague, Czechia
- Århus Universitetshospital, Aarhus, Denmark
- Germany (3):
  - Universitaetsklinikum Heidelberg, Abteilung Neuroonkologie, Heidelberg, Baden-Wurttemberg
  - Klinikum rechts der Isar der TU Muenchen, Neurologische Klinik und Poliklinik, Munich, Bavaria
  - Universitaetsmedizin Rostock, Klinik für Neurologie, Rostock
- Prince of Wales Hospital, Shatin, Hong Kong
- Italy (4):
  - Universitaria Policlinico di Catania, Catania
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Neurological Centre of Latium Dipartimento di Neuroscienze, Rome
- Japan (8):
  - Chiba University Hospital, Chiba, Chiba
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Kyoto Min-iren Chuo Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Kyushu University Hospital, Fukuoka
  - National Center Hospital, NCNP, Tokyo
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- Russia (5):
  - Republican Clinical Hospital for Rehabilitation of Healthcare Ministry of Republic of Tatarstan, Kazan'
  - FSBHI 'Siberian Clinical Center of FMBA', Krasnoyarsk
  - Federal State Budget Institution of Healthcare - Siberian District Medical Center of FMBA of Russia, Novosibirsk
  - SBEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don
  - First Pavlov State Medical University of St.Petersburg, Saint Petersburg
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul University National Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Clinico San Carlos, Madrid
- Cheng Hsin General Hospital, Taipei, Taiwan
- Thailand (3):
  - Navamindradhiraj University, Vajira Hospital, Dusit
  - Thammasat University Hospital, Pathum Thani
  - Sunprasitthiprasong Hospital, Ubon Ratchathani
- Turkey (Türkiye) (6):
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Bilim Universty Medical Fac., Istanbul
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- United Kingdom (2):
  - The Walton Centre, Liverpool
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Pittock SJ, Lennon VA, McKeon A, Mandrekar J, Weinshenker BG, Lucchinetti CF, O'Toole O, Wingerchuk DM. Eculizumab in AQP4-IgG-positive relapsing neuromyelitis optica spectrum disorders: an open-label pilot study. Lancet Neurol. 2013 Jun;12(6):554-62. doi: 10.1016/S1474-4422(13)70076-0. Epub 2013 Apr 26. PMID 23623397
- [Result] Pittock SJ, Berthele A, Fujihara K, Kim HJ, Levy M, Palace J, Nakashima I, Terzi M, Totolyan N, Viswanathan S, Wang KC, Pace A, Fujita KP, Armstrong R, Wingerchuk DM. Eculizumab in Aquaporin-4-Positive Neuromyelitis Optica Spectrum Disorder. N Engl J Med. 2019 Aug 15;381(7):614-625. doi: 10.1056/NEJMoa1900866. Epub 2019 May 3. PMID 31050279
- [Derived] Singh P, Gao X, Kleijn HJ, Bellanti F, Pelto R. Eculizumab Pharmacokinetics and Pharmacodynamics in Patients With Neuromyelitis Optica Spectrum Disorder. Front Neurol. 2021 Nov 3;12:696387. doi: 10.3389/fneur.2021.696387. eCollection 2021. PMID 34803867
- [Derived] Pittock SJ, Fujihara K, Palace J, Berthele A, Kim HJ, Oreja-Guevara C, Nakashima I, Levy M, Shang S, Yountz M, Miller L, Armstrong R, Wingerchuk DM; PREVENT Study Group. Eculizumab monotherapy for NMOSD: Data from PREVENT and its open-label extension. Mult Scler. 2022 Mar;28(3):480-486. doi: 10.1177/13524585211038291. Epub 2021 Sep 9. PMID 34498507
- [Derived] Kim HJ, Nakashima I, Viswanathan S, Wang KC, Shang S, Miller L, Yountz M, Wingerchuk DM, Pittock SJ, Levy M, Berthele A, Totolyan N, Palace J, Barnett MH, Fujihara K; PREVENT Study Group. Eculizumab in Asian patients with anti-aquaporin-IgG-positive neuromyelitis optica spectrum disorder: A subgroup analysis from the randomized phase 3 PREVENT trial and its open-label extension. Mult Scler Relat Disord. 2021 May;50:102849. doi: 10.1016/j.msard.2021.102849. Epub 2021 Feb 20. PMID 33676197
- [Derived] Palace J, Wingerchuk DM, Fujihara K, Berthele A, Oreja-Guevara C, Kim HJ, Nakashima I, Levy M, Terzi M, Totolyan N, Viswanathan S, Wang KC, Pace A, Yountz M, Miller L, Armstrong R, Pittock S; PREVENT Study Group. Benefits of eculizumab in AQP4+ neuromyelitis optica spectrum disorder: Subgroup analyses of the randomized controlled phase 3 PREVENT trial. Mult Scler Relat Disord. 2021 Jan;47:102641. doi: 10.1016/j.msard.2020.102641. Epub 2020 Nov 26. PMID 33310418
- See also: Alexion Clinical Trials Website — http://www.alexionclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Main inclusion criteria were: participants aged ≥ 18 years old with NMO/NMOSD, AQP4 antibody-positive, historical relapse of at least 2 in last 12 months or 3 in last 24 months with at least 1 in 12 months prior to screening, Expanded Disability Status Scale score ≤ 7. If receiving immunosuppressive therapies, must be on a stable maintenance dose.
Groups:
- Eculizumab: Induction Period: Participants received eculizumab (900 milligrams [mg]) via intravenous (IV) infusion once a week (every 7 ± 2 days) for 4 weeks followed by eculizumab 1200 mg for the fifth dose (Week 4).
  Maintenance Period: Participants received eculizumab (1200 mg) via IV infusion every 2 weeks (every 14 ± 2 days) from the sixth dose (Week 6) onwards.
- Placebo: Induction Period: Participants received matching placebo (900 mg) via IV infusion once a week (every 7 ± 2 days) for 4 weeks, followed by matching placebo (1200 mg) for the fifth dose (Week 4).
  Maintenance Period: Participants received matching placebo (1200 mg) via IV infusion every 2 weeks (every 14 ± 2 days) from the sixth dose (Week 6) onwards.
Period: Overall Study
Arm/Group | Eculizumab | Placebo
Started | 96 | 47
Received At Least 1 Dose Of Study Drug (Full Analysis Set (FAS)) | 96 | 47
Completed | 80 | 44
Not Completed | 16 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 12 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who were randomized to treatment and who received at least 1 dose of study drug.
Groups:
- Eculizumab: Induction Period: Participants received eculizumab (900 mg) via IV infusion once a week (every 7 ± 2 days) for 4 weeks followed by eculizumab 1200 mg for the fifth dose (Week 4).
  Maintenance Period: Participants received eculizumab (1200 mg) via IV infusion every 2 weeks (every 14 ± 2 days) from the sixth dose (Week 6) onwards.
- Total: Total of all reporting groups
Arm/Group | Eculizumab | Placebo | Total
Number analyzed (Participants) | 96 | 47 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first dose (years)
  years | 43.9 (13.32) | 45.0 (13.29) | 44.3 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 42 | 130
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 3 | 16
  Not Hispanic or Latino | 78 | 41 | 119
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 37 | 15 | 52
  Black or African American | 9 | 8 | 17
  White | 46 | 24 | 70
  Other or Unknown | 4 | 0 | 4
Overall Stratification Groupings (4 strata) at Randomization [Count of Participants; unit: Participants] — EDSS = Expanded Disability Status Scale; IST = Immunosuppressive Therapy
  High EDSS (≥ 2.5 to ≤ 7): Same IST = High EDSS (≥ 2.5 to ≤ 7) and Continuing on the Same IST(s) since last relapse.
  High EDSS (≥ 2.5 to ≤ 7): Change in IST = High EDSS (≥ 2.5 to ≤ 7) and Changes in IST(s) since last relapse.
  Participants
    Low EDSS (≤ 2.0) | 11 | 5 | 16
    High EDSS (≥ 2.5 to ≤ 7) and Treatment Naive | 12 | 5 | 17
    High EDSS (≥ 2.5 to ≤ 7): Same IST | 44 | 22 | 66
    High EDSS (≥ 2.5 to ≤ 7): Change in IST | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Participants With An Adjudicated On-trial Relapse
Description: An On-trial Relapse was defined as a new onset of neurologic symptoms or worsening of existing neurologic symptoms with an objective change (clinical sign) on neurologic examination that persisted for more than 24 hours as confirmed by the treating physician. An adjudicated On-trial Relapse was defined by the protocol and positively adjudicated by the relapse adjudication committee.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: Full Analysis Set (FAS): all participants who were randomized to treatment, received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
Participants | 3 | 20
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Test type: Other — Treatment Effect; p < 0.0001, Stratified Log-Rank Test; Hazard Ratio (HR) = 0.058, 95% CI 2-sided [0.017 to 0.197] — HR based on a stratified Cox proportional hazards model. Confidence interval = Wald confidence interval. HR for eculizumab compared with placebo represented a 94.2% reduction in the risk of relapse, 95% Wald confidence interval (80.3%, 98.3%)

2. Secondary Outcome: Adjudicated On-trial Annualized Relapse Rate (ARR)
Description: The adjudicated On-trial ARR was computed as the total number of relapses divided by the total number of patient years in the study period. A central independent committee was used to adjudicate all On-trial Relapses as determined by the treating physician. Results reported as adjusted adjudicated On-trial ARR based on a Poisson regression adjusted for randomization strata and historical ARR in 24 months prior to Screening.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: relapses/years on study
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
relapses/years on study | 0.016 [0.005 to 0.050] | 0.350 [0.199 to 0.616]

3. Secondary Outcome: Change From Baseline In EDSS At End Of Study
Description: Disease-related disability was measured by the EDSS. The EDSS is an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. A decrease in score indicates improvement.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
units on a scale | -0.18 (0.814) | 0.12 (0.945)

4. Secondary Outcome: Change From Baseline In Modified Rankin Scale (mRS) Score At End Of Study
Description: Disease-related disability was measured by the mRS score. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered from a neurological disability. The scale ranges from 0 (no disability) to 6 (death) in whole-point increments. A decrease in score indicates improvement.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
units on a scale | -0.2 (0.72) | 0.1 (0.75)

5. Secondary Outcome: Change From Baseline In Hauser Ambulation Index (HAI) Score At End of Study
Description: The HAI evaluates gait and was used to assess the time and effort used by the participant to walk 25 feet (8 meters). The scale ranges from 0 to 9, with 0 being the best score (asymptomatic; fully ambulatory with no assistance) and 9 being the worst (restricted to wheel chair; unable to transfer self independently). A decrease in score indicates improvement.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
units on a scale | -0.4 (1.08) | 0.5 (1.61)

6. Secondary Outcome: Change From Baseline In European Quality Of Life (EuroQoL) Health 5-Dimension Questionnaire (EQ-5D) Visual Analogue Scale At End Of Study
Description: The EuroQoL EQ-5D is a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. Assessments were made using the EQ-5D Visual Analogue Scale, which captures the self-rating of current health status using a visual "thermometer" with the endpoints of 100 (best imaginable health state) at the top and zero (worst imaginable health state) at the bottom. An increase in score indicates improvement.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
units on a scale | 5.4 (18.53) | 0.6 (16.39)

7. Secondary Outcome: Change From Baseline In EuroQoL EQ-5D Index Score At End Of Study
Description: The EuroQoL EQ-5D is a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. Index scores range from less than 0 to 1, with higher scores representing a better health status.
Time Frame: Baseline, Up To 211 Weeks (End of Study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 96 | 47
units on a scale | 0.05 (0.179) | -0.04 (0.212)

ADVERSE EVENTS:
Time Frame: From Day 1 to End of Study (211 Weeks)
Arm/Group | Eculizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/96 | 0/47
Serious Adverse Events (participants affected / at risk) | 30/96 | 26/47
Other Adverse Events (participants affected / at risk) | 86/96 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=96) | Placebo (N=47)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bartholin's abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Renal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 1
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 7 | 16
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Catheterisation venous (Surgical and medical procedures) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Superior mesenteric artery syndrome (Vascular disorders) | 1 | 0
Venous occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=96) | Placebo (N=47)
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 0
Cataract (Eye disorders) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 15 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 16 | 12
Vomiting (Gastrointestinal disorders) | 9 | 8
Asthenia (General disorders) | 5 | 1
Chest discomfort (General disorders) | 2 | 3
Fatigue (General disorders) | 7 | 5
Oedema peripheral (General disorders) | 4 | 3
Pain (General disorders) | 4 | 4
Pyrexia (General disorders) | 6 | 4
Bronchitis (Infections and infestations) | 9 | 2
Conjunctivitis (Infections and infestations) | 9 | 4
Cystitis (Infections and infestations) | 8 | 1
Hordeolum (Infections and infestations) | 7 | 0
Influenza (Infections and infestations) | 11 | 1
Nasopharyngitis (Infections and infestations) | 20 | 9
Pharyngitis (Infections and infestations) | 10 | 3
Pneumonia (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 28 | 6
Urinary tract infection (Infections and infestations) | 11 | 10
Contusion (Injury, poisoning and procedural complications) | 9 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 4
Weight decreased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 10
Dizziness (Nervous system disorders) | 14 | 6
Headache (Nervous system disorders) | 22 | 11
Hypoaesthesia (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 8 | 3
Depression (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 4

LIMITATIONS AND CAVEATS:
After rigorous review of blinded study data, the Sponsor terminated the study at 23 adjudicated events, not the protocol-specified 24. This was not driven by safety or efficacy concerns, but rather by uncertainty in estimating final event occurrence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication rights are tied to the completion of the multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01892345/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01892345/SAP_001.pdf